CLINICAL TRIAL: NCT02612337
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Study of OTO-104 Given as a Single Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: Study of OTO-104 in Subjects With Unilateral Meniere's Disease
Acronym: AVERTS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-201506
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Meniere's Disease
Keywords: Meniere's Disease; Vertigo
MeSH Terms: conditions — Meniere Disease; Vertigo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OTO-104 (Experimental): 12 mg dexamethasone
  Interventions: Drug: OTO-104
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-104 — Single intratympanic injection of 12 mg OTO-104
  Arms: OTO-104
Drug: Placebo — Single intratympanic injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of OTO-104 for the treatment of Meniere's disease.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject has a diagnosis of unilateral Meniere's disease by 1995 American Academy of Otolaryngology - Head and Neck Surgery (AAOHNS) criteria and reports active vertigo for the 2 months prior to the study lead-in period.
* Subject has experienced active vertigo during the lead-in period.
* Subject has documented asymmetric sensorineural hearing loss.
* Subject agrees to maintain their current treatments for Meniere's disease while on-study.

Exclusion Criteria includes, but is not limited to:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has a history of previous endolymphatic sac surgery.
* Subject has a history of previous use of intratympanic (IT) gentamicin in the affected ear.
* Subject has a history of tympanostomy tubes with evidence of perforation or lack of closure.
* Subject has experienced an adverse reaction to IT injection of steroids.
* Subject has used an investigational drug or device in the 3 months prior to screening.
* Subject has previously been randomized to a trial of OTO-104.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Bishop, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Many sites in US. Refer to the contact info listed below., San Diego, California, United States

REFERENCES:
- [Derived] Phillips J, Mikulec AA, Robinson JM, Skarinsky D, Anderson JJ. Efficacy of Intratympanic OTO-104 for the Treatment of Meniere's Disease: The Outcome of Three Randomized, Double-Blind, Placebo-Controlled Studies. Otol Neurotol. 2023 Jul 1;44(6):584-592. doi: 10.1097/MAO.0000000000003886. Epub 2023 Apr 22. PMID 37185596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 166 subjects were randomized and 165 subjects received study drug. The most common reason for screen failure was that there was not a sufficient number of definitive vertigo days in the 28-day lead-in period. The first subject enrolled on October 27, 2015, and the last subject completed the study on July 18, 2017. A total of 47 centers in the US enrolled subjects.
Pre-assignment Details: In addition to meeting all screening visit inclusion criteria, potential subjects had to experience and record at least 4 and a maximum of 22 definitive vertigo day (DVD) during the 4 week lead-in period. In addition, the subject needed to complete at least 22 of 28 diary entries during the 4-week lead-in period. A DVD was defined each day the subject recorded a vertigo episode lasting at least 20 minutes corresponding to a vertigo score of 2 or more.
Period: Overall Study
Arm/Group | OTO-104 | Placebo
Started | 83 | 83
Received Study Drug | 83 | 82
Completed | 80 | 80
Not Completed | 3 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Did not receive study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- OTO-104 (Full Analysis Set): Subjects that were randomized to OTO-104, received study drug, had a baseline definitive vertigo measurement (i.e., at least 1 baseline daily diary entry) for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline (i.e., at least 1 post baseline daily diary entry).
- Placebo (Full Analysis Set): Subjects that were randomized to placebo, received study drug, had a baseline definitive vertigo measurement (i.e., at least 1 baseline daily diary entry) for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline (i.e., at least 1 post baseline daily diary entry).
- Total: Total of all reporting groups
Arm/Group | OTO-104 (Full Analysis Set) | Placebo (Full Analysis Set) | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 61 | 126
  >=65 years | 18 | 21 | 39
Age, Continuous [Median (Full Range); unit: years] | 54.0 [23 to 85] | 58.0 [24 to 83] | 55.7 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 35 | 36 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 73 | 75 | 148
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 74 | 80 | 154
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 83 | 82 | 165
Previous IT Steroid Injection [Count of Participants; unit: Participants] | 20 | 30 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Number of DVD at Week 12 (Defined as the 4-week [28 Days] Interval From Week 9 Through Week 12).
Description: The number of DVDs at Week 12 (defined as the 4-week [28 days] interval from Week 9 through Week 12) was compared between OTO-104 and placebo.
  Week 12 = 12 weeks after dosing at the Baseline visit. Baseline occurred at the end of lead-in and no intervention was administered during lead-in.
Time Frame: Week 12 (3 months)
Population: The full analysis set subjects who were randomized, received study drug, had a baseline definitive vertigo measurement for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline, i.e., at least 1 post-baseline daily diary entry.
Measure: Least Squares Mean (95% Confidence Interval); unit: Definitive Vertigo Day
Arm/Group | OTO-104 (Full Analysis Set) | Placebo (Full Analysis Set)
Number analyzed (Participants) | 83 | 82
Definitive Vertigo Day | 2.191 [1.644 to 2.919] | 2.415 [1.823 to 3.198]
Statistical Analysis 1: Comparison: OTO-104 (Full Analysis Set) vs Placebo (Full Analysis Set); The primary efficacy endpoint was compared between OTO-104 and placebo at the 2-tailed 0.05 alpha level using a generalized Poisson linear mixed model. The model included fixed effects for randomized treatment group, sex, study week, a treatment group by study week interaction, and the count of lead-in period DVD standardized to 28 days as a covariate; Test type: Superiority — The target sample size for each was 160 randomized subjects: 80 in each treatment group stratified by gender. The sample size estimate was chosen to achieve more than 90% power with a significance level of 0.05 2-sided to reject the null hypothesis of no treatment difference for the primary endpoint of DVD; p = 0.623, Regression, Linear; Risk Ratio (RR) = 0.907, 95% CI 2-sided [0.615 to 1.339]

2. Secondary Outcome: Effect of Vertigo on Daily Activities - Number of Days Sick at Home or Bedridden at Week 12 (Month 3)
Description: Questionnaire - subjects were instructed to record the effect on their daily activities of their total vertigo experienced that day using a 5-point scoring system:
  0 = normal activity
  1. = slight limitation
  2. = moderate limitation
  3. = sick at home
  4. = bed ridden
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OTO-104 (Full Analysis Set) | Placebo (Full Analysis Set)
Number analyzed (Participants) | 83 | 82
days | 1.287 (2.8797) | 1.058 (2.077)

3. Secondary Outcome: Otoscopic Examination - Tympanic Membrane Perforation at Week 12 (Month 3)
Description: Otoscopic examinations were conducted at each visit. It was considered important to understand if the tympanic perforation that resulted from the IT injection at the Baseline visit persisted at the end of study visit (Week 12 [Month 3]).
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- OTO-104 (Safety Analysis Set): All subjects who received OTO-104. Subjects were included in this treatment group according to the actual treatment received regardless of their randomized assignment.
- Placebo (Safety Analysis Set): All subjects who received Placebo. Subjects were included in this treatment group according to the actual treatment received regardless of their randomized assignment.
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 82 | 83
participants | 4 | 0

4. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 500 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 500 Hz.
Time Frame: 3 months
Population: Subjects that had no impairment at the Baseline visit (air-bone gap <=10 dB)
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 62 | 70
Participants | 2 | 7

5. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 1000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 1000 Hz.
Time Frame: Week 12 (Month 3)
Population: Subjects that had no impairment at the Baseline visit (air-bone gap <=10 dB
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 70 | 68
Participants | 3 | 3

6. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 2000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 2000 Hz.
Time Frame: Week 12 (Month 3)
Population: Subjects that had no impairment at the Baseline visit (air-bone gap <=10 dB)
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 74 | 78
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Reported or observed during or after dosing with the study drug at the Baseline visit up to the Week 12 (Month 3) end of study visit. The Baseline visit occurred after the Lead-in period when no intervention was administered. Therefore, collection of adverse events started during dosing at the Baseline visit and lasted to the end of the study (Week 12 (Month 3).
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 2/82 | 2/83
Other Adverse Events (participants affected / at risk) | 34/82 | 30/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (Safety Analysis Set) (N=82) | Placebo (Safety Analysis Set) (N=83)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0) — The subject received a dose of study drug and 2 months later underwent a kidney transplant for end-stage renal disease secondary to diabetes after being on a 4-year waiting list. The rejection occurred 2 weeks after that and eventually resolved.
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (Safety Analysis Set) (N=82) | Placebo (Safety Analysis Set) (N=83)
Nasopharyngitis (Infections and infestations) | 3 (3) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 4 (4)
Meniere's disease (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hypoesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT02612337/Prot_SAP_000.pdf